CLINICAL TRIAL: NCT03900559
Title: An Internet-based Treatment for Flying Phobia Using 360º Images: A Feasibility Pilot Study
Brief Title: An Internet-based Treatment for Flying Phobia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: UJaumeI5
Record Dates: First submitted 2019-01-08; First posted 2019-04-03 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Flying Phobia
Keywords: Specific Phobia; Computer-Assisted Exposure; Self-help; Internet-based Therapy; Sense of presence
MeSH Terms: conditions — Aerophobia; Phobia, Specific

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- "NO-FEAR Airlines" program with still images (Experimental): Intervention group that uses "NO-FEAR Airlines" program with still images to carry out the exposure.
  Interventions: Behavioral: NO-FEAR Airlines
- "NO-FEAR Airlines" program with still and navigable images (Experimental): Intervention group that uses "NO-FEAR Airlines" program with still and navigable images to carry out the exposure.
  Interventions: Behavioral: NO-FEAR Airlines
- Waiting list control group (No Intervention): Participants of this group are able to access "NO-FEAR Airlines" program after 6 weeks of waiting period.
  After that period, those participants still interested in receiving assistance are randomly assigned to one of two intervention conditions (only still images or still + navigable images).

INTERVENTIONS:
Behavioral: NO-FEAR Airlines — "NO-FEAR Airlines" is an Internet-based self-applied treatment program that allows people with Flying Phobia the exposure to images and sounds related to their phobic fears on a standard personal computer. The treatment can be totally self-applied.
  "NO-FEAR Airlines" contains 6 scenarios related to the flight process: (1) flight preparation, (2) airport, (3) boarding and taking off, (4) the central part of the flight, (5) the airplane's descent, approach to the runway, and landing, (6) sequences with images and auditory stimuli related to plane crashes.
  Arms: "NO-FEAR Airlines" program with still and navigable images; "NO-FEAR Airlines" program with still images

SUMMARY:
Flying phobia (FP) is one of the most prevalent phobias in our society. However, not all patients benefit from in vivo exposure, given that an important amount of them do not accept the intervention, drop out when they are informed about the intervention procedure, or have problems accessing these therapies.

The aim of the present study is to conduct a feasibility pilot with NO-FEAR Airlines ICBT (Campos et al., 2016) using two types of images in the exposure scenarios (still images vs 360º navigable images). A secondary aim is to explore the potential effectiveness of the two active treatment arms compared to a waiting list control group. Finally, we will explore the role of navigable images compared to the still images in the level of anxiety, sense of presence, and reality judgment in the exposure scenarios and whether the aforementioned variables mediate in treatment efficacy.

Regarding the main aim of this study, we hypothesize that both treatment conditions will be well accepted by the participants, but participants will prefer 360º images over still images.

DETAILED DESCRIPTION:
Flying phobia (FP) is one of the most prevalent phobias in our society. Around 25% of the population that flies experiences intense distress during the flight; around 10% of the general population does not fly due to intense fear and 20% of people depend on alcohol or tranquilizers to overcome the fear of flying.

In vivo exposure is the most effective psychological treatment for specific phobias. However, not all patients benefit from in vivo exposure, given that an important amount of them do not accept the intervention, drop out when they are informed about the intervention procedure, or they have problems to access these therapies.

Information and Communication Technologies (ICTs) can improve treatment adherence and acceptance. Particularly, computerized programs offer remarkable advantages such as a reduction in direct therapeutic contact time, the possibility of standardizing treatment as much as possible with a steep exposure gradient, the low cost and, maybe most importantly, access to patients who would not be very willing to subject themselves to in vivo exposure. The application of cognitive-behavioural procedures such as exposure through interactive computer programs is especially recommended.

On the other hand, it is important to explore the role of the degree of immersion and sense of presence in the psychological treatments with iCBTs due to the contradictory conclusions that had been found in the literature. Therefore, it is expected that the present work advances in the knowledge in this field exploring these factors in an Internet-based self-applied treatment program for FP evaluating if a change in the exposure images used in the program NO-FEAR Airlines (Campos et al., 2016) will be feasible in a future RCT.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18-65 years of age
* To meet current DSM-5 criteria for specific phobia (flying phobia).
* Be willing to participate in the study.
* Be able to use a computer and having an Internet connection.
* Be able to understand and read Spanish.
* Have an e-mail address.

Exclusion Criteria:

* Be receiving psychological treatment for fear of flying.
* A severe mental disorder on Axis I: abuse or dependence of alcohol or other substances, psychotic disorder, dementia, bipolar disorder.
* Severe Personality Disorder.
* Presence of depressive symptomatology, suicidal ideation or plan.
* Presence of heart disease.
* Pregnant women (from the fourth month).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Expectations Scale and Satisfaction Scale (adapted from Borkovec & Nau, 1972) | Up to 12 months
  This self-report inventory measures the patients' expectations before they start the treatment and after they receive a brief explanation about the intervention and their experimental condition. The same questions have to be answered when the patient completes the treatment in order to assess satisfaction. The 6 items are rated from 1 ("Not at all") to 10 ("Highly").
Preferences questionnaire | Up to 12 months
  This questionnaire collects the patient's preferences regarding the two types of images included in this study (navigable and still images) through 5 dichotomous questions where they have to choose one of the two conditions. Participants will answer these questions before the treatment and before knowing the condition to which they are allocated (after the characteristics of each type of image are explained) and after they have completed the treatment (and after seeing a short video showing the image condition they did not receive).
Qualitative Interview | Up to 12 months
  This interview assesses the participant's opinion of the intervention program after finishing it. The interview contains 13 items that the patient has to rate on a scale ranging from 1 ("very little") to 5 ("very much") and explain the reasons for their rating on each question. There are also two open questions where the participants have to give their overall opinion about the intervention program and the program images. In this interview, the perceived sense of presence and reality judgement in each scenario will also be assessed.

SECONDARY OUTCOMES:
Fear and Avoidance Scales (adapted from Marks & Mathews, 1979) | Up to 12 months
  Participants assessed their fear, avoidance and belief in catastrophic thought on a scale ranging from 0 ("No fear at all," "I never avoid") to 10 ("Severe fear," "I always avoid") for situations related with flying.
The Clinician Severity Scale (adapted from Di Nardo, Brown & Barlow, 1994). | Up to 12 months
  The clinician rates the severity of the patient's phobia on a scale from 0 to 8, where 0 = symptom free and 8 = extremely severe.
Patient's Improvement Scale (Adapted from the Clinical Global Impression scale, CGI; Guy, 1976). | Up to 12 months
  One item on the CGI scale was adapted in order to assess the level of improvement achieved by the patient (compared to the baseline) on a 7-point scale (1 "much worse" to 7 "much better"). This scale is answered by the patient.
Fear of Flying Questionnaire (FFQ-II; Bornas et al, 1999) | Up to 12 months
  The FFQ is a 30-item self-report questionnaire that assesses the anxiety the person feels in different situations of the flight process: anxiety during the flight, anxiety experienced getting on the plane, and anxiety experienced due to the observation of neutral or unpleasant flying-related situations. For each item, respondents rate their degree of discomfort associated with the situation on a scale from 1 to 9 (1 = not at all, 9 = very much). Scores range from 30 to 270. Internal consistency was α = .97, and test-retest reliability (15-day retest period) was r = .92 (Bornas et al. 1999).
Fear of Flying Scale (FFS; Haug et al., 1987). | Up to 12 months
  The FFS is a 21-item self-report measure to assess fear in different flying situations. Fear elicited by each situation was rated on a 4-point scale (1= not at all, 4 = very much), with scores ranging from 21 to 84. The original FFS reported a Cronbach's alpha of .94 and retest reliability (after a three-month period) of .86 (Haug et al., 1987).

OTHER OUTCOMES:
Reality Judgement and Presence Questionnaire (RJPQ) (adapted from Baños, Quero, Salvador & Botella, 2007). | Up to 12 months
  This questionnaire is composed by 18 items to assess reality judgment and sense of presence. A 0-10 Likert scale is used to answer all items.
Sense of presence and reality judgment | Up to 12 months
  When the exposure scenario is completed (anxiety level less than 3), the program will assess, on scales from 0 to 10, the extent to which the patients feel present in the situation and the extent to which they feel the situation is real

CONTACTS AND LOCATIONS:
Overall Officials: Soledad Quero, PhD, Study Director — Universitat Jaume I; Cristina Botella, PhD, Study Director — Universitat Jaume I; Sonia Mor, PhD Student, Study Chair — Universitat Jaume I
Locations (1):
- Universitat Jaume I, Castellon, Castellón, Spain

REFERENCES:
- [Background] Botella, C., Osma, J., García-Palacios, A., Quero, S., & Baños, R.M. (2004). Treatment of flying phobia using virtual reality: data from a 1-year follow-up using a multiple baseline design. Clinical Psychology and psychotherapy, 11, 311-323.
- [Background] Campos D, Breton-Lopez J, Botella C, Mira A, Castilla D, Banos R, Tortella-Feliu M, Quero S. An Internet-based treatment for flying phobia (NO-FEAR Airlines): study protocol for a randomized controlled trial. BMC Psychiatry. 2016 Aug 20;16:296. doi: 10.1186/s12888-016-0996-1. PMID 27544428
- [Background] Campos D, Mira A, Breton-Lopez J, Castilla D, Botella C, Banos RM, Quero S. The acceptability of an Internet-based exposure treatment for flying phobia with and without therapist guidance: patients' expectations, satisfaction, treatment preferences, and usability. Neuropsychiatr Dis Treat. 2018 Mar 28;14:879-892. doi: 10.2147/NDT.S153041. eCollection 2018. PMID 29636613
- [Background] Garcia-Palacios A, Botella C, Hoffman H, Fabregat S. Comparing acceptance and refusal rates of virtual reality exposure vs. in vivo exposure by patients with specific phobias. Cyberpsychol Behav. 2007 Oct;10(5):722-4. doi: 10.1089/cpb.2007.9962. PMID 17927544
- [Background] Kazdin, A. E. (2015). Evidence-based psychotherapies II: changes in models of treatment and treatment delivery. South African Journal of Psychology, 45(1), 3-21.
- [Background] Tortella-Feliu M, Botella C, Llabres J, Breton-Lopez JM, del Amo AR, Banos RM, Gelabert JM. Virtual reality versus computer-aided exposure treatments for fear of flying. Behav Modif. 2011 Jan;35(1):3-30. doi: 10.1177/0145445510390801. PMID 21177516
- [Derived] Mor S, Botella C, Campos D, Carlbring P, Tur C, Quero S. An internet-based treatment for flying phobia using 360 degrees images: A feasibility pilot study. Internet Interv. 2022 Feb 16;28:100510. doi: 10.1016/j.invent.2022.100510. eCollection 2022 Apr. PMID 35242593
- [Derived] Mor S, Botella C, Campos D, Tur C, Castilla D, Soler C, Quero S. An Internet-based treatment for Flying Phobia using 360 degrees images: Study protocol for a feasibility pilot study. Internet Interv. 2021 Apr 6;24:100387. doi: 10.1016/j.invent.2021.100387. eCollection 2021 Apr. PMID 33936953